CLINICAL TRIAL: NCT02869646
Title: Acupuncture for PTSD in Combat Veterans
Brief Title: Acupuncture for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Analydata, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLNA-02-15F
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; acupuncture; integrative medicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum acupuncture (Experimental): Traditional Chinese Medicine (TCM) based acupuncture at prescribed sites
  Interventions: Procedure: Procedure: Acupuncture
- Minimal needling (Sham Comparator): shallow and non-acupoint needles at same number of sites
  Interventions: Procedure: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Procedure: Acupuncture — Acupuncture is a general term indicating the insertion and stimulation of needles at one or more prescribed points in order to effect the biology of the individual.
  Other Names: Traditional Chinese Medicine
  Arms: Verum acupuncture
Procedure: Procedure: Sham acupuncture — Sham acupuncture is a general term indicating the use of needles, whether inserted or not, at points on the body that are not expected to have a clinically significant biological effect.
  Other Names: Placebo acupuncture
  Arms: Minimal needling

SUMMARY:
Current treatments for Veterans with PTSD include medications and therapy where the patient talks about traumatic events in order to desensitize to them. While these treatments work for many, a large minority of Veterans do not want medications or exposure therapy. The investigators developed an acupuncture (ACU) treatment for PTSD in order to broaden treatment options. The investigators' first study showed that it helped most people. However, the investigators need better scientific evidence that it works by comparing ACU to a placebo, such as "sham" acupuncture (fewer needles in non-important sites) and determining if ACU alters abnormal physiology in PTSD. In this study 90 Veterans will be randomly assigned (like a coin flip) to receive either ACU or sham. The investigators expect to find that the ACU treated patients have more improvement in PTSD and in physiology (less startle reaction - assessed non-invasively using skin sensors) than the patients in the sham group. This study will provide information to support the use of acupuncture for PTSD at the VA, which will expand treatment options.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is debilitating and common (up to 30% in Vietnam Veterans and 16% in Afghanistan and Iraq Veterans). A significant number of Veterans do not engage in or drop-out from effective trauma-focused therapies due to avoidance from trauma-related memories. Because of this limitation, and because scientific literature suggested that acupuncture might be effective for PTSD symptoms, the investigators developed an acupuncture intervention for PTSD and conducted a clinical trial that showed positive effects. This remains the only high quality trial of acupuncture for PTSD published, because of which the current VA/DoD guidelines for PTSD state that acupuncture is a "B" recommendation (fair evidence, provide service) for PTSD treatment. That civilian study compared acupuncture to an effective therapy (CBT) and a wait-list control, but did not have a placebo control. And, research has shown that Veterans may respond differently to therapies than civilians. More definitive data about the efficacy of acupuncture for PTSD is required in order to recommend it as an "A" evidence-based intervention for PTSD in Veterans. Specifically, it is important to show that acupuncture is better than a placebo control and that it has effects on biological abnormalities of PTSD. The aim of this study is to demonstrate efficacy of acupuncture for PTSD by showing clinical and biological effects that are statistically larger and clinically more important than effects of "sham" acupuncture. Given current knowledge and the need for efficient, ethical and best practices within an experimental design, the primary aim is best accomplished by a randomized controlled trial comparing verum acupuncture (ACU) to placebo minimal needling sham acupuncture (MIN). The goal is to evaluate ACU for a significant positive signal, not to compare ACU to other interventions or to evaluate treatment durability. Acupuncture is delivered in 24 sessions over 12 weeks. The primary hypothesis is that efficacy of ACU for PTSD symptom severity will be large (pre- to post-treatment Cohen's d > 0.8), and significantly better than MIN (between group Cohen's d > 0.30, with 80% probability of detecting a true group difference at p<0.05 (2-sided). The secondary hypothesis is that compared to MIN, ACU will be associated with a significantly larger change from pre- to post-treatment in psychophysiological response (decreased startle by EMG eyeblink during fear conditioning procedure). The study design is a two-arm, parallel-group, prospective randomized controlled trial (RCT). The sample frame is Veterans with chronic PTSD with a sample of convenience from those seeking care at the Long Beach VA. Exclusion criteria are meant to keep out individuals with characteristics that are known to be PTSD treatment confounds, associated with non-adherence or negative response to treatment, that may significantly affect biological assessment, or who may be put at risk of harm. The sample size (90) provides adequate power to test hypotheses. Subjects will be allocated to intervention group by computer-generated adaptive randomization. General linear mixed models will be used to evaluate hypothesized effects over time (mid treatment, end of treatment, 1-month follow-up), controlling for baseline severity of symptoms and demographic characteristics (e.g., age, gender) using intent-to-treat modeling. Outcome effect size (Cohen's d) within and between subjects will be calculated. Interaction terms will be included in the models to evaluate treatment fidelity and treatment expectancy as potential moderators. Study results will provide clinicians and policy makers with more information to make decisions about the rational use of acupuncture for PTSD. This is important because acupuncture is being touted for PTSD by many advocates. It has the potential to reach PTSD sufferers who are not willing to engage in trauma-focused psychotherapy, or for whom current therapies are ineffective. The objective of this project is consistent with priority research areas of specific interest to Clinical Science Research & Development (CSR&D) including PTSD and complementary medicine, and all participants are Veterans at a VA Hospital.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are meant to recruit a relatively homogeneous yet generalizable sample of Veterans with at least moderate chronic PTSD due to combat trauma. Criteria are:

* Veterans age 18 to 55
* DSM-5 criteria for chronic PTSD on the Clinician Administered PTSD Scale (CAPS-5)
* At least moderate PTSD by having a total CAPS-5 score of > 26 and meeting criteria for each of 4 symptom clusters.
* Eligible persons will be allowed to have other symptoms that are commonly comorbid with PTSD. This strategy will provide a feasible and generalizable sample of those with chronic PSTD, but these will not be inclusion or exclusion criteria, e.g.,:

  * anxiety
  * mild to moderate depression
* Women and minorities will be recruited

Exclusion Criteria:

Exclusion criteria are meant to keep out individuals with characteristics that are known to be PTSD treatment confounds, that may significantly affect biological assessment, that indicate past non-adherence or treatment resistance, or who may be put at risk of harm. Criteria are:

* Current and past six-months psychosis
* Substance dependence (evidence of tolerance and/or withdrawal) within the past 6 months
* Thyroid disease
* Decisional incapacity (e.g., dementia)
* Centrally acting medications that have a potential effect on biological expression, e.g.:,

  * beta-blockers
  * opiates
  * >10mg equivalent of diazepam/day
* Pain levels requiring opiate medications
* Known exposure to chemicals or physical trauma that cause neuropsychiatric sequelae
* Severe depression (Beck Depression Inventory-II score >30) that is deemed more clinically significant than PTSD, since this may bias accurate PTSD diagnosis and biological measures
* A diagnosed and untreated sleep breathing disorder (SBD) which is a treatment confound
* A high risk of a SBD as indicated by snoring >50 of nights plus one of:

  * any witnessed apnea
  * feeling non-refreshed in the morning >50 of mornings
  * daytime sleepiness indicated by falling asleep with routine tasks such as watching TV or reading
* Non-response to >2 evidence-based PTSD treatments

  * adequate medication of 12 weeks or completion of Prolonged Exposure (PE)
  * Cognitive Processing Therapy (CPT)
  * or an intensive program
* Treatment non-adherence indicated by stopping treatment or >3 missed appointments in the course of a PTSD Evidenced-Based Treatment (EBT)
* High dissociation as indicated by a score of >25 on the Dissociative Experiences Scale - II (Bernstein & Putnam, 1986)
* Past chronic PTSD prior to military service
* Current active psychotherapy for PTSD
* Having acupuncture in the past year
* Pregnancy
* A person who is on a stable dose (8 weeks) of medication for:

  * depression
  * anxiety
  * PTSD
  * or for sleep, or any other psychoactive medication that may confound the study, and who meet entering criteria and will continue these medications for the duration of the trial will not be excluded (list in Appendix 5)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hollifield, MD, Principal Investigator — VA Long Beach Healthcare System, Long Beach, CA
Locations (1):
- VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollifield M, Hsiao AF, Smith T, Calloway T, Jovanovic T, Smith B, Carrick K, Norrholm SD, Munoz A, Alpert R, Caicedo B, Frousakis N, Cocozza K. Acupuncture for Combat-Related Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Jun 1;81(6):545-554. doi: 10.1001/jamapsychiatry.2023.5651. PMID 38381417
- [Derived] Hollifield M, Hsiao AF, Carrick K, Gory Munoz A, Calloway T, Cocozza K, Smith B, Smith T, Jovanovic T, Norrholm S, Sokhadze E, Reist C. Acupuncture for combat post-traumatic stress disorder: trial development and methodological approach for a randomized controlled clinical trial. Trials. 2021 Sep 6;22(1):594. doi: 10.1186/s13063-021-05394-3. PMID 34488824

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Verum Acupuncture | Minimal Needling
Started | 47 | 45
Completed | 39 | 32
Not Completed | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum Acupuncture | Minimal Needling | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 45 | 92
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 43 | 41 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan Native | 2 | 0 | 2
  Race: White | 23 | 20 | 43
  Race: Asian | 8 | 9 | 17
  Race: Black/African American | 5 | 7 | 12
  Race: More than one | 6 | 9 | 15
  Race: Other | 3 | 0 | 3
Country of Birth [Count of Participants; unit: Participants]
  United States | 35 | 36 | 71
  Other | 12 | 9 | 21
Education Level [Count of Participants; unit: Participants]
  HS/GED | 12 | 7 | 19
  Some College | 18 | 20 | 38
  College Degree | 17 | 18 | 35
Marital Status [Count of Participants; unit: Participants]
  Married | 24 | 21 | 45
  Single | 13 | 7 | 20
  Divorced | 8 | 13 | 21
  Other | 2 | 4 | 6
Religion [Count of Participants; unit: Participants]
  Buddhist | 3 | 1 | 4
  Christian | 22 | 23 | 45
  Muslim | 0 | 2 | 2
  Other | 10 | 11 | 21
  None | 12 | 8 | 20
Annual Income [Count of Participants; unit: Participants]
  Missing | 1 | 0 | 1
  $0 - $19,999 | 3 | 10 | 13
  $20,000 - 34,999 | 6 | 8 | 14
  $35,000 - $49,999 | 13 | 9 | 22
  >$50,000 | 24 | 18 | 42
Employment Status [Count of Participants; unit: Participants]
  Yes | 17 | 24 | 41
  No | 30 | 21 | 51
Combat Exposure [Count of Participants; unit: Participants]
  Light | 1 | 2 | 3
  Moderate Light | 8 | 8 | 16
  Moderate | 16 | 14 | 30
  Moderate Heavy | 14 | 14 | 28
  Heavy | 8 | 7 | 15
Deployment Preparedness [Count of Participants; unit: Participants]
  Low | 4 | 3 | 7
  Moderate | 23 | 22 | 45
  High | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptom Severity on the Clinician Administered PSTD Scale - CAPS 5 From Before to After Treatment
Description: The Clinician Administered PTSD Scale (CAPS) (Blake et al, 1995) is a structured diagnostic interview for PTSD. The CAPS-5 based on DSM-5 criteria will be used. CAPS-5 has 20 symptom items, each rated from 0 (absent) to 4 (severe). A rating of >2 is considered a positive score for diagnostic purposes. The DSM-5 diagnostic rule requires the presence of least one Criterion B symptom, one Criterion C symptom, two Criterion D symptoms, and two Criterion E symptoms in addition to other impairment criteria. The minimum score is 0; the maximum score is 80. A higher score is more severe symptoms and a worse outcome. A DSM-5 CAPS cutoff score of >26 AND meeting each of the 4 symptom cluster criterion will be used for study inclusion and outcomes.
Time Frame: Baseline and 12 weeks
Population: t-tests, statistics of significance and power, and Cohen d tests were used to test hypotheses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Verum Acupuncture | Minimal Needling
Number analyzed (Participants) | 47 | 45
score on a scale | 22.6 (14.1) | 29.1 (11.8)

2. Secondary Outcome: Percentage Change From Baseline in Eyeblink Startle Potentiation
Description: The startle response, measured with electromyography (EMG) of the eyeblink, provides an ideal translational tool to investigate fear conditioning and extinction, since the amygdala is directly connected with the startle circuit. The raw EMG signal will be recorded at a rate of 1000 Hz throughout the experimental session using a 28 Hz high pass and 500 Hz low pass filter (as recommended by guidelines for human eyeblink startle in Blumenthal et al., 2005; Psychophysiology, 42:1-15). Raw signals will be stored and exported for analysis in microvolt ( V) values.
Time Frame: Baseline, 12 weeks
Population: This is only a subset since some either did not participate or dropped out of this component of the research
Measure: Mean (Standard Deviation); unit: % change potentiation of startle
Groups:
- Verum Acupuncture: Real acupuncture per protocol
- Sham Acupuncture: Placebo "minimal" acupuncture
Arm/Group | Verum Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 28 | 26
% change potentiation of startle | -55.8 (21.9) | 6.1 (19.5)

ADVERSE EVENTS:
Time Frame: 16 months
Description: Matches government definitions
Arm/Group | Verum Acupuncture | Minimal Needling
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 21/47 | 16/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum Acupuncture (N=47) | Minimal Needling (N=45)
SAE (General disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Verum Acupuncture (N=47) | Minimal Needling (N=45)
abnormal labs (Blood and lymphatic system disorders) | 7 | 4
Emotional Distress (Nervous system disorders) | 6 | 4
ED visit for pain (Musculoskeletal and connective tissue disorders) | 3 | 0
ED visit other (General disorders) | 2 | 2
General medial symptoms (General disorders) | 9 | 4
PTSD severe related (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02869646/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02869646/SAP_001.pdf